CLINICAL TRIAL: NCT03481270
Title: The Oakland Men's Health Disparities Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marcella Alsan, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 36255
Record Dates: First submitted 2017-10-05; First posted 2018-03-29 (Actual); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Behavior; Cardiovascular Risk Factor; Influenza
MeSH Terms: conditions — Behavior; Influenza, Human

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discordant (Placebo Comparator): Does not receive the concordant provider.
  Interventions: Behavioral: Concordant
- Concordant (Experimental): The intervention is that the subject receives the concordant provider.
  Interventions: Behavioral: Concordant

INTERVENTIONS:
Behavioral: Concordant — We will be randomizing across providers - we are particularly interested in racial concordance.

SUMMARY:
Reducing racial disparities in health outcomes is a major policy concern in the United States. Although there has been recent progress to close the gap, black men continue to experience earlier morbidity and mortality from preventable and manageable medical conditions, and live on average 4.2 years less than their white male peers. An oft-prescribed solution to close this stubborn gap is to increase the diversity of the healthcare workforce. Another common policy tool to increase take-up of preventative healthcare services is financial incentives. In this randomized evaluation, we will estimate the effects of financial incentives and a racially concordant physician on the uptake of preventive health services in Oakland, California.

ELIGIBILITY:
Inclusion Criteria:

* African American male adults

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1374 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbershops / Fleamarkets, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 1374 black men in barbershops and flea markets to take the baseline survey. The subjects were given a coupon which allowed them entrance to the clinic.
Pre-assignment Details: 1374 participants were recruited and completed the baseline survey prior to coming to the clinic. 667 filled out the baseline survey but did not come to the clinic and were not randomized. 70 additional participants were excluded from participation and were not randomized.
Groups:
- Discordant: Subject is not randomized to a concordant provider.
  Concordant: The black male subject is seen by a non-black male doctor.
- Concordant: Subject is randomized to a concordant provider.
  Concordant: The black male subject is seen by a black male doctor.
Period: Overall Study
Arm/Group | Discordant | Concordant
Started | 324 | 313
Completed | 324 | 313
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Numbers are those who presented to the clinic and who met study criteria (African-American, age 18+, male)
Groups:
- Total: Total of all reporting groups
Arm/Group | Discordant | Concordant | Total
Number analyzed (Participants) | 324 | 313 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (16.3) | 42.6 (17.1) | 43.0 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 324 | 313 | 637
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 324 | 313 | 637
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Average education level [Mean (Standard Deviation); unit: score on a scale] — Education level was scored as either zero (less than high school education) or 1 (completed high school education).
  score on a scale | .62 (.49) | .64 (.48) | .63 (.48)

OUTCOME MEASURES:

1. Primary Outcome: Average Take-up of Preventive Services (Post-consultation)
Description: Take-up of preventative services was scored as either zero (did not utilize any post-consultation services) or 1 (utilized at least 1 post-consultation service). Four non-incentivized post-consultation preventive services were offered (for BMI, blood pressure, cholesterol, and/or diabetes); the subject had the opportunity to select service(s) after meeting with their assigned doctor.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Discordant | Concordant
Number analyzed (Participants) | 324 | 313
score on a scale | 0.52 (.36) | .71 (.36)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Discordant | Concordant
All-Cause Mortality (participants affected / at risk) | 0/324 | 0/313
Serious Adverse Events (participants affected / at risk) | 0/324 | 0/313
Other Adverse Events (participants affected / at risk) | 0/324 | 0/313

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT03481270/Prot_SAP_000.pdf